CLINICAL TRIAL: NCT06697717
Title: End-expiratory Transpulmonary Pressure-guided vs EIT-guided PEEP Titration Methods in Patients With Intra-abdominal Hypertension Combined With Acute Respiratory Distress Syndrome: a Randomized Crossover Controlled Study
Brief Title: End-expiratory Transpulmonary Pressure-guided vs Electrical Impedance Tomography-guided PEEP Titration Methods in Patients With Intra-abdominal Hypertension Combined With Acute Respiratory Distress Syndrome: a Randomized Crossover Controlled Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: XiaoJing Zou,MD (Other)
Responsible Party: Sponsor-Investigator, XiaoJing Zou,MD, Clinical Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Organization: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: PEEP20240921
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-01

CONDITIONS: Intra-abdominal Hypertension; Acute Respiratory Distress Syndrome (ARDS)
MeSH Terms: conditions — Intra-Abdominal Hypertension; Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transpulmonary Pressure-Guided PEEP Titration (Experimental)
  Interventions: Other: Transpulmonary Pressure-Guided PEEP Titration in IAH and ARDS Patients
- EIT-Guided PEEP Titration (Experimental)
  Interventions: Other: EIT-Guided PEEP Titration in IAH and ARDS Patients

INTERVENTIONS:
Other: Transpulmonary Pressure-Guided PEEP Titration in IAH and ARDS Patients — After completion of baseline ventilation and lung recruitment, the ventilator was switched to volume-controlled mode, and PEEP was set using an empirical PL-FiO₂ table, with the goal of maintaining end-expiratory transpulmonary pressure (PL) > 0 cmH₂O and end-inspiratory PL ≤ 20 cmH₂O.
  Arms: Transpulmonary Pressure-Guided PEEP Titration
Other: EIT-Guided PEEP Titration in IAH and ARDS Patients — After completion of baseline ventilation and lung recruitment, the ventilator was switched to pressure-controlled mode with a pressure control (PC) of 15 cmH₂O. PEEP was initially set at 35 cmH₂O and then gradually decreased in steps of 3 cmH₂O, with each PEEP level maintained for 2 minutes, down to a minimum of 2 cmH₂O, using the ODCL method for PEEP titration.
  Arms: EIT-Guided PEEP Titration

SUMMARY:
This study aims to adopt a randomized crossover design to compare the effects of end-expiratory transpulmonary pressure-guided PEEP titration and EIT-guided PEEP titration on local lung ventilation, shunt, dead space, and ventilation-perfusion (V/Q) ratio as monitored by EIT. Additionally, it will evaluate their impact on respiratory mechanics, chest wall mechanics, mechanical power, hemodynamics, gas exchange, intra-abdominal pressure, abdominal perfusion pressure, and renal perfusion. By identifying an optimal PEEP titration strategy for patients with intra-abdominal hypertension (IAH) and acute respiratory distress syndrome (ARDS), this study aims to develop a mechanical ventilation approach that maintains lung recruitment and minimizes lung injury while avoiding adverse effects on other organs. The findings could facilitate the clinical application of this strategy and benefit a broader population of patients with IAH and ARDS.

ELIGIBILITY:
Inclusion Criteria:

1. age: 18-80 years;
2. meets IAH ≥12 mmHg;
3. meets the diagnostic criteria of the new global definition of ARDS in the 2023 edition;
4. PaO2/FiO2 ≤ 150;
5. within 36 hours of invasive mechanical ventilation;
6. patients or their family members were consulted, agreed to participate in the trial, and signed an informed consent form.

Exclusion Criteria:

1. Age <18 years or age >80 years;
2. uncorrected shock of any type;
3. chronic obstructive pulmonary disease, interstitial lung disease, pulmonary embolism, right heart failure, pulmonary hypertension, or severe cardiac arrhythmia;
4. pneumothorax or bronchopleural fistula or lobectomy or other surgery of the lungs within 2 weeks of surgery;
5. non-invasive ventilation or transnasal high-flow oxygen;
6. with relevant contraindications to the application of EIT (large chest skin injuries, infections, pacemaker implanters, in vivo automatic defibrillator implantation, etc.) pneumothorax, mediastinal emphysema, massive pleural effusion;
7. oesophageal obstruction, oesophageal perforation, severe oesophageal variceal bleeding, upper gastrointestinal surgery, and other factors that make it impossible to place an oesophageal pressure catheter;
8. diaphragmatic hernia, thoracic deformity; patients with obvious pulmonary hernias;
9. prolongation of prothrombin time (PT), activated partial thromboplastin time (APTT) to two times the high limit of normal values or with active bleeding in the nasopharynx;
10. severe neurological disease: intracranial hypertension or neuromuscular disease, etc;
11. pregnant and lactating women;
12. patients to be treated with ECMO;
13. re-admission to the ICU of patients who have already been included in this study, or who are participating in other clinical studies;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Difference between the optimal PEEP titrated based on end-expiratory transpulmonary pressure and that guided by EIT | After PEEP titration

SECONDARY OUTCOMES:
Electrical impedance tomography (EIT) parameters included: Global inhomogeneity (GI) index、Center of ventilation (CoV)、Shunt fraction、V/Q matching ,and so on | 30-minute ventilation after PEEP titration
Clinical respiratory and hemodynamic parameters | 30-minute ventilation after PEEP titration

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan Union Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No